CLINICAL TRIAL: NCT03571633
Title: A Multicenter, Randomized, Open-label, Phase II Trial Aiming to Evaluate the Impact of Pegfilgrastim on Trastuzumab Anti-tumor Effect and ADCC in Operable HER2 Positive Breast Cancer Patients
Brief Title: Impact of Pegfilgrastim on Trastuzumab Anti-tumor Effect and ADCC in Operable HER2+ Breast Cancer Breast Cancer
Acronym: BREASTIMMU02
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET17-057; 2017-002069-22 (EudraCT Number)
Record Dates: First submitted 2018-06-04; First posted 2018-06-27 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: HER2-positive Breast Cancer; Operable Breast Cancer
Keywords: Pegfilgrastim; Trastuzumab/Paclitaxel; Antibody-dependent cell-mediated cytotoxicity
MeSH Terms: interventions — Trastuzumab; Paclitaxel; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel+Trastuzumab+Pegfilgrastim (Experimental): NEOADJUVANT TREATMENT PERIOD (up to 12 weeks) :Paclitaxel (80 mg/m2, weekly (D1, D8, D15), IV) + Trastuzumab (a loading dose 8 mg/kg at C1D1 followed by 6 mg/kg Q3W, IV OR 600mg, Q3W SC) + Pegfilgrastim (6 mg, Q3W, subcutaneously, the day after the trastuzumab + paclitaxel infusion (i.e. Day 2 of each cycle)).
  ADJUVANT TREATMENT PERIOD (up to 12 months) : Trastuzumab (a loading dose 8 mg/kg at C1D1 followed by 6 mg/kg Q3W, (IV) OR 600mg, Q3W SC)
  Interventions: Drug: Trastuzumab + Paclitaxel; Drug: Pegfilgrastim
- Paclitaxel+Trastuzumab (Active Comparator): NEOADJUVANT TREATMENT PERIOD (up to 12 weeks) :Paclitaxel (80 mg/m2, weekly (D1, D8, D15), IV) + Trastuzumab (a loading dose 8 mg/kg at C1D1 followed by 6 mg/kg Q3W, IV OR 600mg, Q3W SC).
  ADJUVANT TREATMENT PERIOD (up to 12 months) : Trastuzumab (a loading dose 8 mg/kg at C1D1 followed by 6 mg/kg Q3W, (IV) OR 600mg, Q3W SC)
  Interventions: Drug: Trastuzumab + Paclitaxel

INTERVENTIONS:
Drug: Trastuzumab + Paclitaxel — During neoadjuvant period, weekly paclitaxel + trastuzumab (every 3 weeks, Q3W) During adjuvant period, weekly trastuzumab (every 3 weeks, Q3W)
Drug: Pegfilgrastim — During neoadjuvant period, weekly pegfilgrastim (every 3 weeks, Q3W)
  Other Names: Neulasta
  Arms: Paclitaxel+Trastuzumab+Pegfilgrastim

SUMMARY:
First preclinical data suggest that pegfilgrastim could constitute a potent adjuvant for immunotherapy with mAb possessing ADCC/ADCP properties as trastuzumab. Combined treatment of pegfilgrastim and trastuzumab should translate into an increased rate of pathological clinical response. Therefore the investigators' proposal is to evaluate the clinical and biological impact of pegfilgrastim in combination with trastuzumab + paclitaxel in HER2-positive early stage breast cancer patients. Breastimmune02 is a multicenter, randomized, open-label, Phase II trial. Operable HER2+ breast cancer patients previously treated with 4 cycles of standard adriamycine/cyclophosphamide (AC) chemotherapy will be randomized (1:1) to receive in the neoadjuvant setting:Arm A: weekly paclitaxel + trastuzumab (every 3 weeks, Q3W) + pegfilgrastim (Q3W) versus Arm B: weekly paclitaxel + trastuzumab (Q3W).Stratification criteria will be: cN0 versus cN1.

DETAILED DESCRIPTION:
The duration of the neoadjuvant treatment period is planned to be 12 weeks (4 cycles of 3 weeks), except in case of Inacceptable toxicity, or Patient decision, or Withdrawal of consent, or Clinical/radiological signs of disease progression.This neoadjuvant treatment period will be ended with a short term safety visit (STSVNeo) to be scheduled 28 days after the last dose of study treatments (considering the latest study treatments administered). Following the STSVNeo, patients will undergo surgery as per usual practice and pathological response will be centrally assessed by a referent pathologist blinded for the treatment arms.Following surgery, all patients will be treated in the adjuvant setting with trastuzumab administered every 3 weeks for up to 12 months in both arms with clinical assessments every 3 months (cf. Réseau régional de Cancérologie, http://espacecancer.sante-ra.fr/Pages/Accueil.aspx). In case of RH+ disease, endocrine therapy may be initiated as per standard treatment guidelines.This adjuvant treatment period is planned for a maximum of 12 months; except in case of Inacceptable toxicity, or Patient decision, or Withdrawal of consent, or Clinical/radiological signs of disease progression. All randomized and treated patients will be followed-up for relapse and survival for at least 15 months post-randomization (i.e. 1 year post-surgery).

A total of 90 patients will be randomized in the study. (45 per arm). All the data concerning the patients will be recorded in the electronic case report form (eCRF) throughout the study serious adverse event (SAE) reporting will be also paper-based by e-mail and/or Fax. The sponsor will perform the study monitoring and will help the investigators to conduct the study in compliance with the clinical trial protocol, Good Clinical Practices (GCP) and local law requirements

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 years at time of inform consent signature.
* Histologically proven HER2 positive breast cancer defined as 3+ staining intensity by immunohistochemistry (IHC) or a 2+ IHC staining intensity and HER2 gene amplification by FISH.Note: HER2 status will be determined as per institutional practice.
* Operable breast tumor with tumor size and staging: > 20 mm, cN0 or cN1, M0 before any AC or FEC chemotherapy, and at least one measurable lesion ≥10 mm in longest diameter at inclusion according to RECIST 1.1.
* No radiological sign of disease progression at time of randomisation.
* Patient previously treated by 4 cycles of AC or 3 to 4 cycles of FEC without febrile neutropenia and without prior pegfilgrastim treatment.
* Availability of a representative formalin-fixed paraffin-embedded (FFPE) tumor specimen from initial diagnosis (i.e. an archival paraffin block is preferred; or at least 20 unstained slides) with its histological report.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate organ function as defined by the following lab tests (to be carried out within 7 days prior C1D1):Bone marrow (Absolute neutrophil count ≥ 1.5 x 109/L, Platelet count > 100 x 109/L, (without transfusion within 21 days prior to C1D1), Hemoglobin value ≥ 9 g/dL), Renal function (Calculated creatinine clearance by MDRD or CKD-EPI >50 mL/min/1.73m2 or serum creatinine < 1.5ULN), Liver function (Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3ULN, Total serum bilirubin ≤ 1.5 ULN (except for patients with Gilbert disease for whom a total serum bilirubin ≤3 ULN is acceptable), Coagulation (INR and aPTT≤ 1.5 ULN)
* Adequate cardiac function with Mean resting corrected QT interval (QTc), calculated using Fridericia's formula, ≤470ms obtained from 3 electrocardiograms (ECGs) and Systolic blood pressure <160mmHg and Diastolic blood pressure <100mmHg (hypertension controlled by standard medical treatment is allowed)
* Women of childbearing potential (entering the study after a confirmed menstrual period and who have a negative pregnancy test within 7 days before C1D1) must agree to use two methods of medically acceptable forms of contraception from the date of negative pregnancy test to 3 months after the last study drug intake
* Patients should be able and willing to comply with study visits and procedures as per protocol
* Patients should understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed.
* Patients must be covered by a medical insurance.

Exclusion Criteria:

* Patients with inflammatory breast cancer.
* Previous exposure to pegfilgrastim or trastuzumab. Note: the use of filgrastim (non pegylated form only) is authorized prior to the randomisation.
* Patients requiring the concomitant use of any forbidden treatment including: Any other anti-cancer treatments not listed in the protocol, including chemotherapy, radiotherapy, immunotherapy, targeted therapy or biologic therapy for cancer treatment, Any investigational treatment.
* Any contra-indication to trastuzumab, paclitaxel, and pegfilgrastim respective SPCs including:Hypersensitivity to trastuzumab, murine proteins, or to any of the excipients listed in trastuzumab SPC, Severe dyspnea at rest due to complications of advanced malignancy or requiring supplementary oxygen therapy, Hypersensitivity to pegfilgrastim or filgrastim, or to any of the excipients listed in SPC, Hereditary problems of fructose intolerance, Hypersensitivity to paclitaxel or to any excipient, particularly macrogolglycerol ricinoleate, Patients with history of or active cardiac disease including myocardial infarction (MI), angina pectoris requiring medical treatment, congestive heart failure NYHA (New York Heart Association) Class ≥II, other cardiomyopathy, cardiac arrhythmia requiring medical treatment, clinically significant cardiac valvular disease, and hemodynamic effective pericardial effusion.
* Active secondary malignancy unless this malignancy is not expected to interfere with the evaluation of study endpoints and is approved by the sponsor. Examples of the latter include basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix. Patients with a completely treated prior malignancy and no evidence of disease for ≥ 2 years are eligible.
* Pregnant or breast-feeding female patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | 16 weeks after start of treatment
  Defined as ypT0 ypN0 or ypT0/is ypN0 after 12 weeks of treatment by trastuzumab + paclitaxel ± pegfilgrastim with ypT0/Tis ypN0 defined as absence of invasive cancer in the breast and axillary nodes in all surgically excised specimens.

SECONDARY OUTCOMES:
Disease Free survival | At least 15 months following randomisation
  From the date of randomisation until the date of event defined as the first documented relapse after surgery or death from any cause.
Time to relapse | At least 15 months following randomisation
  From the time of treatment start until the first documented relapse
Overall survival | At least 15 months following randomisation
  From the date of randomisation to the date of death from any cause
Adverse events reporting | At least 15 months following randomisation
  Based mainly on the frequency of AE graded according to the common toxicity criteria grading system (CTCAE-V4.03).

OTHER OUTCOMES:
Trastuzumab ADCC activity | At Baseline, at Day 1 of Cycle 2 (each cycle is a 21-day cycle) and at surgery
  Analysis of the levels of the ADCC tumor samples
HER2 signaling | At Baseline, at Day 1 of Cycle 2 (each cycle is a 21-day cycle) and at surgery
  Evaluation of the levels of phosphorylated components of PI3K/mTOR and Ras/Raf /MAPK signaling (IHC or IF)
Immune effector cells activity | At Baseline, at Day 1 of Cycle 2 (each cycle is a 21-day cycle) and at surgery
  Analysis of activity of immune effector cells (frequency, function, activation status and ADCC)
TGFbeta levels | At Baseline
  Levels of TGFβ (bioactive and non-bioactive) in serum, plasma and platelets
Residual disease of class | At surgery
  Evaluation of RCB Class by local pathologist and blinded independent central review after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Olivier TREDAN, MD, Principal Investigator — Centre Leon Berard
Locations (9):
- France (9):
  - Institut Sainte Catherine, Avignon
  - CHRU Besançon, Besançon
  - Centre de Lutte contre le Cancer Jean Perrin, Clermont-Ferrand
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Centre Leon Berard, Lyon
  - Hopital Prive Jean Mermoz, Lyon
  - Centre Hospitalier Annecy Genevois, Pringy
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne
  - Clinique Charcot, Sainte-Foy-lès-Lyon

REFERENCES:
- [Background] Ferlay J, Shin HR, Bray F, Forman D, Mathers C, Parkin DM. Estimates of worldwide burden of cancer in 2008: GLOBOCAN 2008. Int J Cancer. 2010 Dec 15;127(12):2893-917. doi: 10.1002/ijc.25516. PMID 21351269
- [Background] Wolff AC, Hammond ME, Hicks DG, Dowsett M, McShane LM, Allison KH, Allred DC, Bartlett JM, Bilous M, Fitzgibbons P, Hanna W, Jenkins RB, Mangu PB, Paik S, Perez EA, Press MF, Spears PA, Vance GH, Viale G, Hayes DF; American Society of Clinical Oncology; College of American Pathologists. Recommendations for human epidermal growth factor receptor 2 testing in breast cancer: American Society of Clinical Oncology/College of American Pathologists clinical practice guideline update. J Clin Oncol. 2013 Nov 1;31(31):3997-4013. doi: 10.1200/JCO.2013.50.9984. Epub 2013 Oct 7. PMID 24101045
- [Background] Wolff AC, Hammond ME, Schwartz JN, Hagerty KL, Allred DC, Cote RJ, Dowsett M, Fitzgibbons PL, Hanna WM, Langer A, McShane LM, Paik S, Pegram MD, Perez EA, Press MF, Rhodes A, Sturgeon C, Taube SE, Tubbs R, Vance GH, van de Vijver M, Wheeler TM, Hayes DF; American Society of Clinical Oncology/College of American Pathologists. American Society of Clinical Oncology/College of American Pathologists guideline recommendations for human epidermal growth factor receptor 2 testing in breast cancer. Arch Pathol Lab Med. 2007;131(1):18-43. doi: 10.5858/2007-131-18-ASOCCO. PMID 19548375
- [Background] Zhou BP, Hung MC. Dysregulation of cellular signaling by HER2/neu in breast cancer. Semin Oncol. 2003 Oct;30(5 Suppl 16):38-48. doi: 10.1053/j.seminoncol.2003.08.006. PMID 14613025
- [Background] Slamon D, Eiermann W, Robert N, Pienkowski T, Martin M, Press M, Mackey J, Glaspy J, Chan A, Pawlicki M, Pinter T, Valero V, Liu MC, Sauter G, von Minckwitz G, Visco F, Bee V, Buyse M, Bendahmane B, Tabah-Fisch I, Lindsay MA, Riva A, Crown J; Breast Cancer International Research Group. Adjuvant trastuzumab in HER2-positive breast cancer. N Engl J Med. 2011 Oct 6;365(14):1273-83. doi: 10.1056/NEJMoa0910383. PMID 21991949
- [Background] Untch M, Rezai M, Loibl S, Fasching PA, Huober J, Tesch H, Bauerfeind I, Hilfrich J, Eidtmann H, Gerber B, Hanusch C, Kuhn T, du Bois A, Blohmer JU, Thomssen C, Dan Costa S, Jackisch C, Kaufmann M, Mehta K, von Minckwitz G. Neoadjuvant treatment with trastuzumab in HER2-positive breast cancer: results from the GeparQuattro study. J Clin Oncol. 2010 Apr 20;28(12):2024-31. doi: 10.1200/JCO.2009.23.8451. Epub 2010 Mar 22. PMID 20308670
- [Background] Gianni L, Eiermann W, Semiglazov V, Manikhas A, Lluch A, Tjulandin S, Zambetti M, Vazquez F, Byakhow M, Lichinitser M, Climent MA, Ciruelos E, Ojeda B, Mansutti M, Bozhok A, Baronio R, Feyereislova A, Barton C, Valagussa P, Baselga J. Neoadjuvant chemotherapy with trastuzumab followed by adjuvant trastuzumab versus neoadjuvant chemotherapy alone, in patients with HER2-positive locally advanced breast cancer (the NOAH trial): a randomised controlled superiority trial with a parallel HER2-negative cohort. Lancet. 2010 Jan 30;375(9712):377-84. doi: 10.1016/S0140-6736(09)61964-4. PMID 20113825
- [Background] Gianni L, Eiermann W, Semiglazov V, Lluch A, Tjulandin S, Zambetti M, Moliterni A, Vazquez F, Byakhov MJ, Lichinitser M, Climent MA, Ciruelos E, Ojeda B, Mansutti M, Bozhok A, Magazzu D, Heinzmann D, Steinseifer J, Valagussa P, Baselga J. Neoadjuvant and adjuvant trastuzumab in patients with HER2-positive locally advanced breast cancer (NOAH): follow-up of a randomised controlled superiority trial with a parallel HER2-negative cohort. Lancet Oncol. 2014 May;15(6):640-7. doi: 10.1016/S1470-2045(14)70080-4. Epub 2014 Mar 20. PMID 24657003
- [Background] Kute T, Stehle JR Jr, Ornelles D, Walker N, Delbono O, Vaughn JP. Understanding key assay parameters that affect measurements of trastuzumab-mediated ADCC against Her2 positive breast cancer cells. Oncoimmunology. 2012 Sep 1;1(6):810-821. doi: 10.4161/onci.20447. PMID 23162748
- [Background] Deauvieau F, Ollion V, Doffin AC, Achard C, Fonteneau JF, Verronese E, Durand I, Ghittoni R, Marvel J, Dezutter-Dambuyant C, Walzer T, Vie H, Perrot I, Goutagny N, Caux C, Valladeau-Guilemond J. Human natural killer cells promote cross-presentation of tumor cell-derived antigens by dendritic cells. Int J Cancer. 2015 Mar 1;136(5):1085-94. doi: 10.1002/ijc.29087. Epub 2014 Aug 6. PMID 25046660
- [Background] Hernandez-Ilizaliturri FJ, Jupudy V, Ostberg J, Oflazoglu E, Huberman A, Repasky E, Czuczman MS. Neutrophils contribute to the biological antitumor activity of rituximab in a non-Hodgkin's lymphoma severe combined immunodeficiency mouse model. Clin Cancer Res. 2003 Dec 1;9(16 Pt 1):5866-73. PMID 14676108
- [Background] Cornet S, Mathe D, Chettab K, Evesque A, Matera EL, Tredan O, Dumontet C. Pegfilgrastim Enhances the Antitumor Effect of Therapeutic Monoclonal Antibodies. Mol Cancer Ther. 2016 Jun;15(6):1238-47. doi: 10.1158/1535-7163.MCT-15-0759. Epub 2016 Mar 17. PMID 26988998
- [Background] Cartron G, Zhao-Yang L, Baudard M, Kanouni T, Rouille V, Quittet P, Klein B, Rossi JF. Granulocyte-macrophage colony-stimulating factor potentiates rituximab in patients with relapsed follicular lymphoma: results of a phase II study. J Clin Oncol. 2008 Jun 1;26(16):2725-31. doi: 10.1200/JCO.2007.13.7729. Epub 2008 Apr 21. PMID 18427151
- [Background] Bossuyt V, Provenzano E, Symmans WF, Boughey JC, Coles C, Curigliano G, Dixon JM, Esserman LJ, Fastner G, Kuehn T, Peintinger F, von Minckwitz G, White J, Yang W, Badve S, Denkert C, MacGrogan G, Penault-Llorca F, Viale G, Cameron D; Breast International Group-North American Breast Cancer Group (BIG-NABCG) collaboration. Recommendations for standardized pathological characterization of residual disease for neoadjuvant clinical trials of breast cancer by the BIG-NABCG collaboration. Ann Oncol. 2015 Jul;26(7):1280-91. doi: 10.1093/annonc/mdv161. Epub 2015 May 27. PMID 26019189
- [Background] Lin Y, Kikuchi S, Obata Y, Yagyu K; Tokyo Research Group on Prevention of Gastric Cancer. Serum levels of transforming growth factor beta1 are significantly correlated with venous invasion in patients with gastric cancer. J Gastroenterol Hepatol. 2006 Feb;21(2):432-7. doi: 10.1111/j.1440-1746.2005.03939.x. PMID 16509870
- [Background] Tas F, Yasasever CT, Karabulut S, Tastekin D, Duranyildiz D. Serum transforming growth factor-beta1 levels may have predictive and prognostic roles in patients with gastric cancer. Tumour Biol. 2015 Mar;36(3):2097-103. doi: 10.1007/s13277-014-2817-9. Epub 2014 Nov 13. PMID 25391430
- [Background] Lin Y, Kikuchi S, Tamakoshi A, Obata Y, Yagyu K, Inaba Y, Kurosawa M, Kawamura T, Motohashi Y, Ishibashi T; JACC Study Group. Serum transforming growth factor-beta1 levels and pancreatic cancer risk: a nested case-control study (Japan). Cancer Causes Control. 2006 Oct;17(8):1077-82. doi: 10.1007/s10552-006-0048-0. PMID 16933058
- [Background] Zhao J, Liang Y, Yin Q, Liu S, Wang Q, Tang Y, Cao C. Clinical and prognostic significance of serum transforming growth factor-beta1 levels in patients with pancreatic ductal adenocarcinoma. Braz J Med Biol Res. 2016 Jul 25;49(8):e5485. doi: 10.1590/1414-431X20165485. PMID 27464025
- [Background] Tas F, Karabulut S, Yasasever CT, Duranyildiz D. Serum transforming growth factor-beta 1 (TGF-beta1) levels have diagnostic, predictive, and possible prognostic roles in patients with melanoma. Tumour Biol. 2014 Jul;35(7):7233-7. doi: 10.1007/s13277-014-1984-z. Epub 2014 Apr 27. PMID 24771267
- [Background] Xu S, Yang S, Sun G, Huang W, Zhang Y. Transforming growth factor-beta polymorphisms and serum level in the development of osteosarcoma. DNA Cell Biol. 2014 Nov;33(11):802-6. doi: 10.1089/dna.2014.2527. Epub 2014 Aug 6. PMID 25098449